CLINICAL TRIAL: NCT04815811
Title: Study of the Sex Differences in Inflammatory Diseases in Children
Acronym: SepsiX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Collaborators: Belgium Kid's Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P2019/LABO/SepsiX
Record Dates: First submitted 2020-10-21; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2020-10

CONDITIONS: Sex Differences in Immune Response; Acute Inflammatory Diseases in Children
Keywords: Sex, immunology, inflammation, child, sepsis, UTI, pneumonia
MeSH Terms: conditions — Coitus; Inflammation; Sepsis; Urinary Tract Infections; Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children suffering from acute inflammatory processes. (Experimental): The study population will consist of male and female children, aged from 6 months to 7 years old, admitted to the hospital for one of the three following types of acute inflammatory processes:
  * Urinary tract infection caused by Escherichia coli
  * Pneumonia with pleural effusion caused by Streptococcus pneumoniae
  * Sepsis
  Interventions: Other: Blood collection; Other: Stool collection
- Control group (Other): Male and female children, aged from 6 months to 7 years old, admitted to the hospital for a scheduled operation for a non-inflammatory pathology.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood samples collections to evaluation of the potential role of the sex chromosomes in the innate immune response by analyzing inflammatory cytokine production (IL-1β, IL-6, IL-8, IL-10, TNF-α and IFN-α), studying the cell diapedesis receptor CD99 on PMNs, monocytes, and lymphocytes, analyzing the contribution of X-linked genes of the TLR pathways and the influence of X-linked miRNAs.
Other: Stool collection — Fecal sample collection to delineate microbiome contribution, we will study the gut microbiota in faecal samples obtained from the recruited patients.
  Arms: Children suffering from acute inflammatory processes.

SUMMARY:
Sexual differences in innate immune response have been demonstrated and were mainly attributed to the influence of the sex steroids (1-18). However, recent clinical data revealed significant differences in inflammatory markers between boys and girls suffering from acute and chronic inflammatory diseases (19-23). Sex hormone levels in prepubertal children are particularly low and insufficient to explain the gender differences observed in inflammatory conditions from neonates to the elderly, suggesting the contribution of another mechanism, such as the influence of genes situated on the sex chromosomes and involved in the inflammatory response.

The aim of this work is to evaluate the role of the X chromosome in the sex differences in inflammatory diseases in children. In order to discriminate more precisely the role of the X chromosome relatively to the sex steroids in the sex-specific inflammatory response, some innate immune functions related to X-linked genes will be evaluated in whole blood from prepubertal children of both sexes, suffering from acute inflammatory processes such as pyelonephritis caused by Escherichia coli, pneumonia with pleural effusion caused by Streptococcus pneumoniae or sepsis

DETAILED DESCRIPTION:
Many studies demonstrated immune differences between men and women suffering from acute and chronic inflammatory processes. In cases of acute inflammatory diseases, such as sepsis, females have better prognosis comparing to males (1,24-28).

On the contrary, worse prognosis for women is observed in chronic inflammatory diseases such as asthma or cystic fibrosis (8-10,12,13,29).

Sex-depended inflammatory response was attributed to the influence of sex hormones on the immune system. (2,15-18). However recent studies revealed differences in the clinical outcome but also in inflammatory markers between boys and girls suffering from acute and chronic inflammatory diseases (19-23). Sex hormone levels in prepubertal children are particularly low and insufficient to explain the gender differences observed in inflammatory conditions from neonates to the elderly, suggesting the contribution of another mechanism, such as the influence of genes situated on the sex chromosomes and involved in the inflammatory response.

The aim of this work is to identify the potential X-linked mechanisms responsible for some of the differences between boys and girls in the inflammatory response, making the girls more at risk of developing complications in chronic inflammatory diseases and the boys more at risk of lethal complications in severe acute inflammatory diseases like sepsis. Several genes coding for innate immunity components are linked to the X chromosome such as diapedesis molecule CD99 or TLR pathway proteins genes. (30-33). X chromosome is also highly enriched in genes encoding micro RNAs (miRNAs) involved in the post-transcriptional regulation of gene expression which play a critical role in immune inflammatory response (34-36).

Thus, in order to discriminate more precisely the role of the X chromosome relatively to the sex steroids in the sex-specific inflammatory response, some innate immune functions related to X-linked genes will be evaluated in whole blood from prepubertal children of both sexes, suffering from acute inflammatory processes such as pyelonephritis caused by Escherichia coli, pneumonia with pleural effusion caused by Streptococcus pneumoniae or sepsis. We will also study the correlations between inflammatory and clinical markers of the disease activity to identify prognosis indicators depending on the sex. Additionally, to delineate microbiome contribution, we will study the gut microbiota in stool samples obtained from the recruited patients.

ELIGIBILITY:
Inclusion Criteria of Experimental group :

* Male (XY) and female (XX) aged from 6 months to 7 years old.
* Subject hospitalized either for:

  (1) Urinary tract infection caused by Escherichia Coli, with:
* Temperature ≥ to 38,5°C
* Urinalysis

  * Leukocyte esterase +
  * AND/OR Nitrites +
  * AND/OR pyuria (≥ 100WBC/mm³)
  * AND/OR bacteriuria.
* Urinalysis

  * Clean catch voided urine: > 10^4 Escherichia Coli colony form unit (CFU)/mm (urine collection method for children >3 years old or toilet trained children or by stimulation for children <3 years old)
  * Transurethral bladder catheterisation: > 10^4 Escherichia Coli colony form unit (CFU)/mm³ (urine collection method for children <3 years old).
  * Suprapubic aspiration: > 1 Escherichia Coli colony form unit (CFU)/mm³ (urine collection method for children <3 years old).

    (2) Pneumonia with pleural effusion with :
* Temperature ≥ 38,5°C
* Chest radiography/ultrasound: Pleural effusion
* Streptococcus pneumoniae identified on blood or pleural fluid culture or by PCR

  (3) Sepsis with:
* Documented or suspected infection
* Temperature < 36° or > 38.3°C
* Heart rhythm:

  * 2 SD above normal for age
  * 6-23 months: >180/min
  * 24-71 months: >140/min
  * 72-84 months: >130/min
* Respiratory Rate:

  * 6-23 months: >35/min
  * 24 - 71 months: >30/min
  * 72-84 months: >20/min
* WBC:

  * 6-23 months: >17500/µL or <5000/µL
  * 24-71 months: >15500/µL or <6000/µL
  * 72-84 months: >13500/µL or <4500/µL
  * and/or CRP (blood) > 2SD above normal
* And at least two of the following:

  * PaO2/FiO2 <300
  * Proven need for >50% FiO2 to maintain saturation ≥ 92%
  * Need for mechanical ventilation
  * Glasgow score < 11
  * Urine output < 0,5mL/kg/h for at least 2h
  * Creatinine:

    * 6-11 months: >0,4mg/dL
    * 12-23 months: >0,5mg/dL
    * 24-59 months: >0,8mg/dL
    * 60-84 months: >1mg/dL
    * Or creatinine increase more than 0,5 mg/dL
  * Platelet count <100000/mL
  * Bilirubin >2 mg/dL
  * Mean arterial pressure (MAP)

    * 6-11 months: <55 mmHg
    * 12 -23 months: <60 mmHg
    * 24-59 months: <62 mmHg
    * 60-84 months: <65 mmHg
  * SBP less than two SD below normal for age
  * Prolonged capillary refill: > 5 sec

Inclusion Criteria of Control group :

* Male (XY) and female (XX) aged from 6 months to 7 years old.
* Scheduled surgical intervention for a non-infectious pathology.

Exclusion Criteria:

* Use of antithrombotic drugs (acetylsalicylic acid, thienopyridines, dipyridamol, glycoprotein IIb / IIIa antagonists, vitamin K antagonists, heparins).
* Congenital or acquired immunodeficiency: immunosuppressive drugs, hematopoietic stem cells transplantation, immunoglobulin therapy, extracorporeal membrane oxygenation (ECMO).
* Hemodialysis.
* 48h following cardiac operation of any type.
* Malignant cancer.
* HIV.

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — equity between male and female among the sample size
Enrollment: 160 (Estimated)
Dates: Start 2019-08-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole blood production of cytokine IL-6 | within 24 hours of hospital admission (Day 0)
  The production of IL6 is measured by multiplex techniques.

SECONDARY OUTCOMES:
Whole blood production of cytokine IL-1β | within 24 hours of hospital admission (Day 0)
Whole blood production of cytokine IL-8 | within 24 hours of hospital admission (Day 0)
Whole blood production of cytokine IL-10 | within 24 hours of hospital admission (Day 0)
Whole blood production of cytokine TNF-α | within 24 hours of hospital admission (Day 0)
Whole blood production of cytokine interferon-α | within 24 hours of hospital admission (Day 0)
Intracellular quantity of the phosphorylated forms of NF-κB p65 in leukocyte population. | within 24 hours of hospital admission (Day 0)
Intracellular quantity of the phosphorylated forms of ERK1/2 in leukocyte population. | within 24 hours of hospital admission (Day 0)
Intracellular quantity of the phosphorylated forms of p38 MAPK in leukocyte population. | within 24 hours of hospital admission (Day 0)
Expression of the cell diapedesis receptor CD99 on PMNs | within 24 hours of hospital admission (Day 0)
  Measurements of cell diapedesis receptor CD99 on leukocytes will be performed by flow cytometry
Expression of the cell diapedesis receptor CD99 on monocytes | within 24 hours of hospital admission (Day 0)
  Measurements of cell diapedesis receptor CD99 on leukocytes will be performed by flow cytometry
Expression of the cell diapedesis receptor CD99 on lymphocytes | within 24 hours of hospital admission (Day 0)
  Measurements of cell diapedesis receptor CD99 on leukocytes will be performed by flow cytometry
Expression of TLR2 on PMNs | within 24 hours of hospital admission (Day 0)
  Measurements of intracellular phosphorylated forms of TLR pathway proteins as well as the expression of TLR2 and TLR4 will be performed by flow cytometry
Expression of TLR2 on monocytes | within 24 hours of hospital admission (Day 0)
  Measurements of intracellular phosphorylated forms of TLR pathway proteins as well as the expression of TLR2 and TLR4 will be performed by flow cytometry
Expression of TLR2 on lymphocytes | within 24 hours of hospital admission (Day 0)
  Measurements of intracellular phosphorylated forms of TLR pathway proteins as well as the expression of TLR2 and TLR4 will be performed by flow cytometry
Expression of TLR4 on PMNs | within 24 hours of hospital admission (Day 0)
  Measurements of intracellular phosphorylated forms of TLR pathway proteins as well as the expression of TLR2 and TLR4 will be performed by flow cytometry
Expression of TLR4 on monocytes | within 24 hours of hospital admission (Day 0)
  Measurements of intracellular phosphorylated forms of TLR pathway proteins as well as the expression of TLR2 and TLR4 will be performed by flow cytometry
Expression of TLR4 on lymphocytes | within 24 hours of hospital admission (Day 0)
  Measurements of intracellular phosphorylated forms of TLR pathway proteins as well as the expression of TLR2 and TLR4 will be performed by flow cytometry
BTK gene expression | within 24 hours of hospital admission (Day 0)
  Measurements will be performed using the Quantitect Reverse Transcription Kit (Qiagen, Manchester, UK) for quantitative PCR (qPCR) on leucocytes.
IRAK1 gene expression | within 24 hours of hospital admission (Day 0)
  Measurements will be performed using the Quantitect Reverse Transcription Kit (Qiagen, Manchester, UK) for quantitative PCR (qPCR) on leucocytes.
NEMO gene expression | within 24 hours of hospital admission (Day 0)
  Measurements will be performed using the Quantitect Reverse Transcription Kit (Qiagen, Manchester, UK) for quantitative PCR (qPCR) on leucocytes.
Expression of X-linked miRNAs in leucocytes | within 24 hours of hospital admission (Day 0)
  Expression of X-linked miRNAs is measured by sequencing and qRT-PCR on leucocytes and/or plasma samples.
Expression of X-linked miRNAs in plasma | within 24 hours of hospital admission (Day 0)
  Expression of X-linked miRNAs is measured by sequencing and qRT-PCR on leucocytes and/or plasma samples.
Leukocyte population | within 24 hours of hospital admission (Day 0)
  White blood cell count including neutrophils, monocytes, monocytes subtypes and lymphocytes.
Leukocyte population | Day 1
  White blood cell count including neutrophils, monocytes, monocytes subtypes and lymphocytes. Only applicable for the sepsis sub-group
Leukocyte population | Day 2
  White blood cell count including neutrophils, monocytes, monocytes subtypes and lymphocytes. Only applicable for the sepsis sub-group
Leukocyte population | Day 3
  White blood cell count including neutrophils, monocytes, monocytes subtypes and lymphocytes. Only applicable for the sepsis sub-group
CRP | within 24 hours of hospital admission (Day 0)
CRP | Day 1
  Only applicable for the sepsis sub-group
CRP | Day 2
  Only applicable for the sepsis sub-group
CRP | Day 3
  Only applicable for the sepsis sub-group
Total 17β-estradiol | within 24 hours of hospital admission (Day 0)
Testosterone | within 24 hours of hospital admission (Day 0)
IGF1 | within 24 hours of hospital admission (Day 0)
Microbiome analysis | During subject hospitalisation
pSOFA score | within 24 hours of hospital admission (Day 0)
  Only applicable for the sepsis sub-group. The pSOFA will be evaluated every 24 hours in order to compare laboratory and clinical data. The score will be based on the PaO2: FiO2 or SpO2: FiO2 ratio, the platelet count, the bilirubin level, the Mean Arterial Pressure (MAP), the Glasgow score and the creatinine level.
pSOFA score | Day 1
  Only applicable for the sepsis sub-group. The pSOFA will be evaluated every 24 hours in order to compare laboratory and clinical data. The score will be based on the PaO2: FiO2 or SpO2: FiO2 ratio, the platelet count, the bilirubin level, the Mean Arterial Pressure (MAP), the Glasgow score and the creatinine level.
pSOFA score | Day 2
  Only applicable for the sepsis sub-group. The pSOFA will be evaluated every 24 hours in order to compare laboratory and clinical data. The score will be based on the PaO2: FiO2 or SpO2: FiO2 ratio, the platelet count, the bilirubin level, the Mean Arterial Pressure (MAP), the Glasgow score and the creatinine level.
pSOFA score | Day 3
  Only applicable for the sepsis sub-group. The pSOFA will be evaluated every 24 hours in order to compare laboratory and clinical data. The score will be based on the PaO2: FiO2 or SpO2: FiO2 ratio, the platelet count, the bilirubin level, the Mean Arterial Pressure (MAP), the Glasgow score and the creatinine level.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Popotals, MD, Principal Investigator — HUDERF
Locations (1):
- HUDERF, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schroder J, Kahlke V, Staubach KH, Zabel P, Stuber F. Gender differences in human sepsis. Arch Surg. 1998 Nov;133(11):1200-5. doi: 10.1001/archsurg.133.11.1200. PMID 9820351
- [Background] Angele MK, Pratschke S, Hubbard WJ, Chaudry IH. Gender differences in sepsis: cardiovascular and immunological aspects. Virulence. 2014 Jan 1;5(1):12-9. doi: 10.4161/viru.26982. Epub 2013 Nov 5. PMID 24193307
- [Background] Wichmann MW, Inthorn D, Andress HJ, Schildberg FW. Incidence and mortality of severe sepsis in surgical intensive care patients: the influence of patient gender on disease process and outcome. Intensive Care Med. 2000 Feb;26(2):167-72. doi: 10.1007/s001340050041. PMID 10784304
- [Background] Schoeneberg C, Kauther MD, Hussmann B, Keitel J, Schmitz D, Lendemans S. Gender-specific differences in severely injured patients between 2002 and 2011: data analysis with matched-pair analysis. Crit Care. 2013 Nov 29;17(6):R277. doi: 10.1186/cc13132. PMID 24289182
- [Background] Moss M, Mannino DM. Race and gender differences in acute respiratory distress syndrome deaths in the United States: an analysis of multiple-cause mortality data (1979- 1996). Crit Care Med. 2002 Aug;30(8):1679-85. doi: 10.1097/00003246-200208000-00001. PMID 12163776
- [Background] Carr MJ, Moss E, Waters A, Dean J, Jin L, Coughlan S, Connell J, Hall WW, Hassan J. Molecular epidemiological evaluation of the recent resurgence in mumps virus infections in Ireland. J Clin Microbiol. 2010 Sep;48(9):3288-94. doi: 10.1128/JCM.00434-10. Epub 2010 Jul 21. PMID 20660212
- [Background] McClelland EE, Smith JM. Gender specific differences in the immune response to infection. Arch Immunol Ther Exp (Warsz). 2011 Jun;59(3):203-13. doi: 10.1007/s00005-011-0124-3. Epub 2011 Mar 26. PMID 21442309
- [Background] Vink NM, Postma DS, Schouten JP, Rosmalen JG, Boezen HM. Gender differences in asthma development and remission during transition through puberty: the TRacking Adolescents' Individual Lives Survey (TRAILS) study. J Allergy Clin Immunol. 2010 Sep;126(3):498-504.e1-6. doi: 10.1016/j.jaci.2010.06.018. PMID 20816186
- [Background] Venn A, Lewis S, Cooper M, Hill J, Britton J. Questionnaire study of effect of sex and age on the prevalence of wheeze and asthma in adolescence. BMJ. 1998 Jun 27;316(7149):1945-6. doi: 10.1136/bmj.316.7149.1945. No abstract available. PMID 9641931
- [Background] Chen W, Mempel M, Schober W, Behrendt H, Ring J. Gender difference, sex hormones, and immediate type hypersensitivity reactions. Allergy. 2008 Nov;63(11):1418-27. doi: 10.1111/j.1398-9995.2008.01880.x. PMID 18925878
- [Background] Raghavan D, Varkey A, Bartter T. Chronic obstructive pulmonary disease: the impact of gender. Curr Opin Pulm Med. 2017 Mar;23(2):117-123. doi: 10.1097/MCP.0000000000000353. PMID 27977622
- [Background] Fogarty A, Hubbard R, Britton J. International comparison of median age at death from cystic fibrosis. Chest. 2000 Jun;117(6):1656-60. doi: 10.1378/chest.117.6.1656. PMID 10858398
- [Background] Sweezey NB, Ratjen F. The cystic fibrosis gender gap: potential roles of estrogen. Pediatr Pulmonol. 2014 Apr;49(4):309-17. doi: 10.1002/ppul.22967. Epub 2013 Dec 11. PMID 24339235
- [Background] Betteridge JD, Armbruster SP, Maydonovitch C, Veerappan GR. Inflammatory bowel disease prevalence by age, gender, race, and geographic location in the U.S. military health care population. Inflamm Bowel Dis. 2013 Jun;19(7):1421-7. doi: 10.1097/MIB.0b013e318281334d. PMID 23518811
- [Background] Ahmed SA, Talal N. Sex hormones and the immune system--Part 2. Animal data. Baillieres Clin Rheumatol. 1990 Apr;4(1):13-31. doi: 10.1016/s0950-3579(05)80241-9. PMID 2282659
- [Background] Lahita RG. Sex hormones and the immune system--Part 1. Human data. Baillieres Clin Rheumatol. 1990 Apr;4(1):1-12. doi: 10.1016/s0950-3579(05)80240-7. No abstract available. PMID 2282655
- [Background] Bouman A, Heineman MJ, Faas MM. Sex hormones and the immune response in humans. Hum Reprod Update. 2005 Jul-Aug;11(4):411-23. doi: 10.1093/humupd/dmi008. Epub 2005 Apr 7. PMID 15817524
- [Background] Bosch F, Angele MK, Chaudry IH. Gender differences in trauma, shock and sepsis. Mil Med Res. 2018 Oct 26;5(1):35. doi: 10.1186/s40779-018-0182-5. PMID 30360757
- [Background] Casimir GJ, Heldenbergh F, Hanssens L, Mulier S, Heinrichs C, Lefevre N, Desir J, Corazza F, Duchateau J. Gender differences and inflammation: an in vitro model of blood cells stimulation in prepubescent children. J Inflamm (Lond). 2010 Jun 2;7:28. doi: 10.1186/1476-9255-7-28. PMID 20525175
- [Background] Casimir GJ, Mulier S, Hanssens L, Knoop C, Ferster A, Hofman B, Duchateau J. Chronic inflammatory diseases in children are more severe in girls. Shock. 2010 Jul;34(1):23-6. doi: 10.1097/SHK.0b013e3181ce2c3d. PMID 20016408
- [Background] Casimir GJ, Mulier S, Hanssens L, Zylberberg K, Duchateau J. Gender differences in inflammatory markers in children. Shock. 2010 Mar;33(3):258-62. doi: 10.1097/SHK.0b013e3181b2b36b. PMID 19543152
- [Background] Casimir GJ, Lefevre N, Corazza F, Duchateau J. Sex and inflammation in respiratory diseases: a clinical viewpoint. Biol Sex Differ. 2013 Sep 1;4:16. doi: 10.1186/2042-6410-4-16. eCollection 2013. PMID 24128344
- [Background] Lefevre N, Noyon B, Biarent D, Corazza F, Duchateau J, Casimir G. Sex Differences in Inflammatory Response and Acid-Base Balance in Prepubertal Children with Severe Sepsis. Shock. 2017 Apr;47(4):422-428. doi: 10.1097/SHK.0000000000000773. PMID 27755508
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Wichmann et al. - 2000 - Incidence and mortality of severe sepsis in surgic.pdf [Internet]. [cited 2019 Feb 27]. Available from: https://link.springer.com/content/pdf/10.1007/s001340050041.pdf
- [Background] The effect of sex on asthma control from the National Asthma Survey - Journal of Allergy and Clinical Immunology [Internet]. [cited 2019 Feb 27]. Available from: https://www.jacionline.org/article/S0091-6749(08)02373-7/fulltext
- [Background] Johnston CM, Lovell FL, Leongamornlert DA, Stranger BE, Dermitzakis ET, Ross MT. Large-scale population study of human cell lines indicates that dosage compensation is virtually complete. PLoS Genet. 2008 Jan;4(1):e9. doi: 10.1371/journal.pgen.0040009. Epub 2007 Dec 13. PMID 18208332
- [Background] Lefevre N, Corazza F, Duchateau J, Desir J, Casimir G. Sex differences in inflammatory cytokines and CD99 expression following in vitro lipopolysaccharide stimulation. Shock. 2012 Jul;38(1):37-42. doi: 10.1097/SHK.0b013e3182571e46. PMID 22575993
- [Background] Spolarics Z. The X-files of inflammation: cellular mosaicism of X-linked polymorphic genes and the female advantage in the host response to injury and infection. Shock. 2007 Jun;27(6):597-604. doi: 10.1097/SHK.0b013e31802e40bd. PMID 17505297
- [Background] Li Q, Verma IM. NF-kappaB regulation in the immune system. Nat Rev Immunol. 2002 Oct;2(10):725-34. doi: 10.1038/nri910. PMID 12360211
- [Background] O'Connell RM, Rao DS, Chaudhuri AA, Baltimore D. Physiological and pathological roles for microRNAs in the immune system. Nat Rev Immunol. 2010 Feb;10(2):111-22. doi: 10.1038/nri2708. PMID 20098459
- [Background] Ceribelli A, Satoh M, Chan EK. MicroRNAs and autoimmunity. Curr Opin Immunol. 2012 Dec;24(6):686-91. doi: 10.1016/j.coi.2012.07.011. Epub 2012 Aug 14. PMID 22902047
- [Background] Dorhoi A, Iannaccone M, Farinacci M, Fae KC, Schreiber J, Moura-Alves P, Nouailles G, Mollenkopf HJ, Oberbeck-Muller D, Jorg S, Heinemann E, Hahnke K, Lowe D, Del Nonno F, Goletti D, Capparelli R, Kaufmann SH. MicroRNA-223 controls susceptibility to tuberculosis by regulating lung neutrophil recruitment. J Clin Invest. 2013 Nov;123(11):4836-48. doi: 10.1172/JCI67604. PMID 24084739
- [Background] Morgan E, Varro R, Sepulveda H, Ember JA, Apgar J, Wilson J, Lowe L, Chen R, Shivraj L, Agadir A, Campos R, Ernst D, Gaur A. Cytometric bead array: a multiplexed assay platform with applications in various areas of biology. Clin Immunol. 2004 Mar;110(3):252-66. doi: 10.1016/j.clim.2003.11.017. PMID 15047203
- [Background] Kuczynski J, Stombaugh J, Walters WA, Gonzalez A, Caporaso JG, Knight R. Using QIIME to analyze 16S rRNA gene sequences from microbial communities. Curr Protoc Bioinformatics. 2011 Dec;Chapter 10:10.7.1-10.7.20. doi: 10.1002/0471250953.bi1007s36. PMID 22161565